CLINICAL TRIAL: NCT01067885
Title: MARIS - Prospective, Multicenter Registry
Brief Title: A Post-market Registry of the MARIS-stent (Invatec) Implanted in the Superficial Femoral Artery
Acronym: MARIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Care Center Prof. Mathey, Prof. Schofer, Ltd. (Other)
Collaborators: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MARIS-01
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Peripheral Artery Disease
Keywords: Nitinol Stent; Superficial femoral artery; SFA; Angioplasty; peripheral artery disease; peripheral artery obstructive disease; PAOD; PAD; Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MARIS-stent (Invatec) — stenting of SFA with Maris nitinol stent/s
  Other Names: Maris nitinol stent (Invatec, Italy)

SUMMARY:
The MARIS Register is a prospective, multicenter registry of implantation in the superficial femoral artery (SFA) with a CE marked stent (Maris / Invatec) intended to capture initial angiographic success, complication rate and symptomatic related revascularization by following the clinical process and duplex examinations at 6 and 12 month.

DETAILED DESCRIPTION:
Recent data suggest that there is some evidence for a reduced restenosis rate for the implantation of a self expanding nitinol stent in the superficial femoral artery (SFA) compared to implantation of balloon expandable stents or single balloon inflation (ABSOLUTE study/FAST study).

The purpose of the Maris Register is to evaluate the primary nitinol stent implantation in an all comer population with diseased SFA.

The MARIS Register is a prospective, multicenter registry of the implantation of at least one at most five nitinol stents (Maris / Invatec) in the SFA without limitations for stenosis or occlusion length.

The registry includes 998 patients from 13 German investigational sites. Clinical data are captured on electronic case report forms

The primary endpoint is the target lesion revascularization after 12 month

Secondary endpoints are :

* Restenosis rate > 50% according to ultrasound criteria
* Restenosis rate > 70% according to ultrasound criteria
* Location of restenosis (proximal, middle, distal AFS)
* Number of stent fractures (grading according to FESTO criteria)
* Procedure related complication rate
* Vascular complication rate within 12 month
* Amputations within 12 month
* Deaths within 12 month

In order to measure the restenosis the peak systolic velocity (PSV) is to be measured in two sections during the duplex ultrasound examinations at 6 and 12 month. First measurement is performed 2cm proximal to the first stent, second measurement at the location where the maximum peak velocity over all lesions/all implanted stents is measured.

The clinical status includes the patient´s Fontaine classification.

ELIGIBILITY:
Inclusion criteria

* stent implantation in SFA is possible
* existing SFA stenosis 70-100 % (visual estimation)
* absence of homodynamically relevant stenosis in A. poplitea
* at least one lower limb run off vessel

Exclusion criteria

* pregnancy
* life expectancy less than 1 year
* coagulation disorder
* chronic anticoagulation therapy
* active gastrointestinal bleeding
* thrombolytic therapy within 72 hours before intervention
* hyperthyreosis
* severe contrast agent allergy
* allergy to concomittant medication
* severe liver disease
* thrombus in target lesion
* target lesion extend into A. poplitea
* severe calcification of target vessel, where no successful pre-dilatation is feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1051 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
target lesion revascularization | 1 year

SECONDARY OUTCOMES:
Restenosis rate > 50% according to ultrasound criteria | 6 and 12 month
Restenosis rate > 70% according to ultrasound criteria | 6 and 12 month
Location of restenosis (proximal, middle, distal AFS) | 6 and 12 month
Number of stent fractures (grading according to FESTO criteria) | 12 month
Procedure related complication rate | Discharge
Vascular complication rate within 12 month | 12month
Amputations within 12 month | 12month
Deaths within 12 month | 12month

CONTACTS AND LOCATIONS:
Overall Officials: Hans Krankenbeg, MD, Principal Investigator — MCC Prof. Mathey, Prof. Schofer

REFERENCES:
- [Derived] Krankenberg H, Tubler T, Sixt S, Fischer M, Schmiedel R, Schulte KL, Balzer JO, Kieback A, Fiehn E, Wittenberg G, Ali T, Tiefenbacher C, Jahnke T, Steinkamp HJ, Wegscheider K, Treszl A, Ingwersen M, Zeller T. German multicenter real-world registry of stenting for superficial femoral artery disease: clinical results and predictive factors for revascularization. J Endovasc Ther. 2014 Aug;21(4):463-71. doi: 10.1583/13-4625R.1. PMID 25101571